CLINICAL TRIAL: NCT04150133
Title: The Effects and Tolerability of a Prescribed Low Residue Diet the Day Before Colonoscopy on the Cleanliness of the Colon vs. the Traditional Clear Liquid, Day Before Diet With the Use of the Clenpiq Bowel Purgative
Brief Title: Effects and Tolerability With Clenpiq and Low Residue Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillmont GI (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: foodprep2019
Record Dates: First submitted 2019-10-24; First posted 2019-11-04 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Colonoscopy Preparation
Keywords: low residue diet

STUDY DESIGN:
Intervention Model Description: single blind trial of FDA approved preparation with per labeling clear liquid diet versus a single day low residue diet
Who Masked: Investigator
Masking Description: Investigator will be ignorant of how preparation was taken
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Clear Liquid Arm (Active Comparator): Following instructions with FDA-labeled clear liquids
  Interventions: Other: Low Residue Diet
- Low Residue Diet Arm (Experimental): Following instructions for a low residue diet along with FDA-labeled clear liquids
  Interventions: Other: Low Residue Diet

INTERVENTIONS:
Other: Low Residue Diet — Variable cohort will eat 3 low residue meals on the day prior to their planned colonoscopy

SUMMARY:
The Efficacy of Clenpiq utilized per FDA labeling, with a low residue diet the day before colonoscopy.

DETAILED DESCRIPTION:
This study proposes to assess the use of a low residue diet of a prescribed nature the day before colonoscopy for breakfast, lunch and early dinner. Clinical outcomes utilizing the low residue diet will be compared to the Food and Drug Administration (FDA) approved split dose labeling, including the traditional clear liquid diet the day before colonoscopy utilizing the Clenpiq (Ferring Pharmaceuticals) bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects age 18-80 requiring colonoscopy for appropriate indications

Exclusion Criteria:

* Active diarrhea (Greater than 3 unformed stools daily)
* Constipation (Less than 3 spontaneous bowel movements per week) Each within 2 weeks of the scheduled Colonoscopy.

Additional exclusion criteria would include;

* Subjects with a history of inflammatory bowel disease
* Colonic resection of any length
* Pregnant women
* American Society of Anesthesiologists (ASA) score greater than 3
* Body Mass Index (BMI) greater than 50
* Previous reaction to this bowel preparation or contraindications to taking Clenpiq per the package labeling guidelines.
* Subjects unable to give their own informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Statistical equivalence of the clear liquid and low residue cohorts | During Colonoscopy Up to 24 hours
  Using the Boston Bowel Preparation Score, the 3 sections of the colon will be graded on adequacy of preparation at the colonoscopy

SECONDARY OUTCOMES:
Polyp Detection Rate | Post Procedure Up to 24 hours
  Number of polyps detected and removed per total number of patients in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Bertiger, MD, Principal Investigator — Hillmont GI
Locations (1):
- Hillmont GI, Flourtown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No